CLINICAL TRIAL: NCT03798002
Title: Effects of Neuro-muscular Exercise Training Verses Isolated Quadriceps Training Program in Patients With Mild to Moderate Knee Osteoarthritis
Brief Title: Neuro-muscular Exercise Training Verses Quadriceps Training in Mild to Moderate Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RiphahI Maryam Khan
Record Dates: First submitted 2019-01-05; First posted 2019-01-09 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Knee Osteoarthritis
Keywords: isolated quadriceps training; Neuro-muscular exercise training; knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuro-muscular exercise training Group (Experimental): Neuro-muscular exercise training will be administer to Knee OA patients.
  Interventions: Other: Neuro-muscular exercise training Group
- quadriceps training program (Active Comparator): quadriceps stretching and strengthening exercises will be administer to Knee OA patients.
  Interventions: Other: quadriceps training program

INTERVENTIONS:
Other: Neuro-muscular exercise training Group — Training takes place 3 days a week for 8 weeks follow up, under the supervision of physical therapist A training session lasts for 40 minutes, and consists of three parts.
  PART 1:Warming up:
  warm-up period consists of ergometer cycling for 10 minutes
  PART 2: Circuit program:
  comprises four exercises, core stability/postural function; postural orientation; lower extremity muscle strength; and functional exercises. Each exercise is performed 2-3 sets 10-15 repetitions.
  PART 3:Cooling down:
  The cooling down part consists of walking exercises forward and backwards, about 10 meters in each direction, in front of mirror (mobility exercises for the lower extremity muscles for a total of about 10 minutes. Changes in patient's symptom assessed by structural questionnaire
  Arms: Neuro-muscular exercise training Group
Other: quadriceps training program — Apply Tens (10min+ hot pack 7-10min) Before excercise ROM,Quadriceps and hamstring stretching exercise's and strengthening exercises.
  4th-6th week (in addition): Straight leg raise, Quads over a roll, Hamstring curls. 7th and 8th week (in addition): Elastic band exercise, Hamstring curls, Quads chair, isometric strengthening All exercises are performed in set of 10 repetitions. 1 set of all exercises was twice a day for first 3 week, and 2 sets twice a day until 6th week and then 3 sets twice a day until 8th week
  Arms: quadriceps training program

SUMMARY:
A randomized controlled trial in which Neuro-muscular exercise training and Isolated quadriceps training program would be applied on patients with symptomatic knee Osteoarthritis by using different tools and changes would be examined pre and post intervention .The participants fulfilling inclusion criteria would be randomly allocated to two groups. Both groups received different protocols and will be assessed on data collection tool on their first and last visit by using Numeric Pain Rating Scale (NPRS), The Western Ontario and McMaster Osteoarthritis Index (WOMAC), Timed Up and Go test (TUG test), 30sec chair stand test,6min walk test (6MWT).Participants of both groups will be pre-tested before the application of interventional programs and post-tested after the application of respective intervention.

DETAILED DESCRIPTION:
The knee joint is a complex modified hinge joint with the greatest range of movement. Three bones come together to form the joint, which are the femur, tibia, and patella. Osteoarthritis, commonly known as wear-and-tear arthritis, is a condition in which the natural cushioning between joints, cartilage wears away. The bones of the joints rub more closely against one another with less of the shock-absorbing benefits of cartilage. The rubbing results in pain, swelling, stiffness, decreased ability to move and, sometimes, the formation of bone spurs.

Osteoarthritis is widespread among physically active individuals . The quadriceps weakness commonly associated with osteoarthritis of the knee is widely believed to result from disuse atrophy secondary to pain in the involved joint. However, quadriceps weakness may be an etiologic factor in the development of osteoarthritis. Several studies have indicated that Physical modalities for the treatment of knee pain in patients with osteoarthritis include physical therapy, exercise, weight loss, and the use of braces or heel wedges. High- and low-intensity aerobic exercises are equally effective in improving functional status, gait, pain, and aerobic capacity in persons with knee osteoarthritis water-based and land-based exercises reduce knee pain and physical disability and aerobic walking, quadriceps strengthening, resistance exercise reduce pain and disability.Several proptocols are available for management of knee joint osteoarthritis. These protocols include Neuro motor training exercise and isolated quadriceps training program. Neuromotor training is basically combination of three parts warming up, a circuit program, and cooling down. Main principle of Neuro-motor training is to improve sensorimotor control and compensatory functional stability.[3]Patients with symptomatic osteoarthritis pain, stiffness, flexibility and decreases range of motion is a common clinical finding. Flexibility is an important component of fitness needed for most desirable musculoskeletal functioning and maximizing the performance of physical activities. Flexibility is a biomechanical property of the body tissues and it determines the range of motion possible without injury at a joint or group of joints. Decrease range of motion has been shown to predispose a person to several musculoskeletal overuse injuries and considerably affect a person level of function.Changes in joint appearance/ joint deformities be one of the more commonly established causes of osteoarthritis. The target in treating patients with OA should be the safest possible intervention, with the best pain relief and prevention of further functional disability. Neuromotor training is also one of the treatment option related to physical therapy in reducing knee pain with home plane exercises to gain required ROM and resume function. Time up and go test (TUG test).the tug is internationally accepted functional dynamic test of balance with known reliability and validity as well as being low cost and easy to apply. The tug test measures the time in seconds that takes a subject to stand up from chair and sit down. Subject will score less than 10 seconds are consider normal, less than 15 sec are at risk of fall ,less than 20 sec are independent in ambulation and able to climb the stairs, and greater than 30 seconds need help with chair. The 30 Second Chair Stand Test, in conjunction with other measures such as the 4-Stage Balance Test, Timed Up and Go (TUG) Test and an assessment of postural hypotension can help to indicate if a patient is at risk of falling. Purpose is to test leg strength and endurance Equipment: A chair with a straight back, without arm rests, placed against a wall to prevent it moving. Sit in the middle of the chair. Place each hand on the opposite shoulder crossed at the wrists. Place your feet flat on the floor. Keep your back straight and keep your arms against your chest. On "Go", rise to a full standing position and then sit back down again. Repeat this for 30 seconds. On "Go" begin timing. Do not continue if you feel the patient may fall during the test. Count the number of times the patient comes to a full standing position in 30 seconds and record it in the box below. If the patient is over halfway to a standing position when 30 seconds have elapsed, count it as a stand. If the patient must use his or her arms to stand then stop the test and record "0" for the number below.The western Ontario and McMaster universities osteoarthritis (womac) is a widely used by health professionals to evaluate the condition of patient with osteoarthritis of knee . womac measures 5 items for pain score 0-20. 2 for stiffness score 0-8 and 17 for functional limitation score 0-68. Physical functioning question of daily activities such as siting standing walking lying on bed taking of socks getting in or out of bath. Numeric pain rating scale (NPRs) is used for measure of pain intensity. In NPRS 0-10 integers that best reflects the intensity of pain. 0 represent no pain.

Previous studies were more focused on hydrotherapeutic exercises, muscle stretching strengthening, aerobics. There is still a challenge to explore best type of exercise therapy for improving sensorimotor function, alleviating symptoms and showing the disease process in different sub groups of patients with degenerative knee disease

ELIGIBILITY:
Inclusion Criteria:

* UL/BL knee OA,
* Age 40-65, both genders,
* American college of rheumatology criteria for knee OA,
* Grade 2 or 3 on Kellgren/Lawrence classification for Knee OA.

Exclusion Criteria:

* Knee surgery
* Rheumatoid arthritis
* Any neurological condition affecting lower limbs and balance
* Use of assistive devices for walking.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
WOMAC Scale | From baseline to 8th week
  WOMAC is western Onterio and McMaster Osteoarthritis Index. Its scores are from 0-100

SECONDARY OUTCOMES:
Numeric pain rating scale(NPRS) | From baseline to 8th week
  Numeric pain rating scale is used to measure pain. Its score is from 0-10, with 0 means no pain and10 means worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: imran Amjad, Phd*, Principal Investigator — Associate Professor
Locations (2):
- Pakistan (2):
  - Imran Amjad, Islamabad, Punjab Province
  - Riphah International University, Islamabad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weng MC, Lee CL, Chen CH, Hsu JJ, Lee WD, Huang MH, Chen TW. Effects of different stretching techniques on the outcomes of isokinetic exercise in patients with knee osteoarthritis. Kaohsiung J Med Sci. 2009 Jun;25(6):306-15. doi: 10.1016/S1607-551X(09)70521-2. PMID 19560995
- [Background] Slemenda C, Brandt KD, Heilman DK, Mazzuca S, Braunstein EM, Katz BP, Wolinsky FD. Quadriceps weakness and osteoarthritis of the knee. Ann Intern Med. 1997 Jul 15;127(2):97-104. doi: 10.7326/0003-4819-127-2-199707150-00001. PMID 9230035
- [Background] Bhatia D, Bejarano T, Novo M. Current interventions in the management of knee osteoarthritis. J Pharm Bioallied Sci. 2013 Jan;5(1):30-8. doi: 10.4103/0975-7406.106561. PMID 23559821
- [Background] Merashly M, Uthman I. Management of knee osteoarthritis: an evidence-based review of treatment options. J Med Liban. 2012 Oct-Dec;60(4):237-42. PMID 23461090
- [Background] Holsgaard-Larsen A, Clausen B, Sondergaard J, Christensen R, Andriacchi TP, Roos EM. The effect of instruction in analgesic use compared with neuromuscular exercise on knee-joint load in patients with knee osteoarthritis: a randomized, single-blind, controlled trial. Osteoarthritis Cartilage. 2017 Apr;25(4):470-480. doi: 10.1016/j.joca.2016.10.022. Epub 2016 Nov 9. PMID 27836677
- [Background] Villadsen A, Overgaard S, Holsgaard-Larsen A, Christensen R, Roos EM. Immediate efficacy of neuromuscular exercise in patients with severe osteoarthritis of the hip or knee: a secondary analysis from a randomized controlled trial. J Rheumatol. 2014 Jul;41(7):1385-94. doi: 10.3899/jrheum.130642. Epub 2014 Jun 15. PMID 24931956
- [Background] Ageberg E, Nilsdotter A, Kosek E, Roos EM. Effects of neuromuscular training (NEMEX-TJR) on patient-reported outcomes and physical function in severe primary hip or knee osteoarthritis: a controlled before-and-after study. BMC Musculoskelet Disord. 2013 Aug 8;14:232. doi: 10.1186/1471-2474-14-232. PMID 23924144
- [Background] Bennell KL, Egerton T, Wrigley TV, Hodges PW, Hunt M, Roos EM, Kyriakides M, Metcalf B, Forbes A, Ageberg E, Hinman RS. Comparison of neuromuscular and quadriceps strengthening exercise in the treatment of varus malaligned knees with medial knee osteoarthritis: a randomised controlled trial protocol. BMC Musculoskelet Disord. 2011 Dec 5;12:276. doi: 10.1186/1471-2474-12-276. PMID 22141334